CLINICAL TRIAL: NCT04270175
Title: Daratumumab, Pomalidomide, and Dexamethasone (DPd) in Relapsed/Refractory Light Chain Amyloidosis Patients Previously Exposed to Daratumumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-12021159
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Amyloid; AL Amyloidosis; Refractory AL Amyloidosis
MeSH Terms: conditions — Alzheimer Disease; Immunoglobulin Light-chain Amyloidosis | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- daratumumab/pomalidomide/dexamethasone (Experimental): Pomalidomide:
  (4mg orally) on days 1-21 of a 28-day cycle
  Dexamethasone:
  * 20mg IV as premedication on days 1, 8, 15, and 22
  * 20mg orally the day after daratumumab dosing for cycles 1-2 of induction
  * 40mg IV as premedication on days 1 and 15 on daratumumab treatment days
  * 40mg orally on non-daratumumab days (8 and 15) for cycles 3-6
  * 20mg on day 1 of every cycle as premedication on daratumumab dosing day 1 in maintenance cycles (cycles 7 and beyond)
    * If you are a subject age 70 and older, the dexamethasone dosing will be reduced by 50% at the time of induction.
  Daratumumab:
  * 1800mg sub-cutaneously weekly x8 weeks
  * 1800mg sub-cutaneously every 2 weeks during induction (cycles 3-6)
  * 1800mg sub-cutaneously every 4 weeks cycles 7 and beyond
  Interventions: Drug: Daratumumab SC; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab SC — Given as 1800mg via injection
  Other Names: Faspro
Drug: Pomalidomide — Given as 4mg oral capsule
Drug: Dexamethasone — Given as 20mg or 40 mg IV and 20mg or 40mg oral tablet.

SUMMARY:
This study will test the hypothesis that in patients with previous daratumumab exposure, combination therapy of daratumumab, pomalidomide, and dexamethasone (DPd) will yield higher complete remission (CR) rates in relapsed/refractory amyloidosis than historical pomalidomide/dexamethasone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary AL amyloidosis of tissue
* Relapsed and/or refractory AL amyloidosis
* Has received daratumumab or Faspro in any prior line of therapy
* Prior pomalidomide exposure allowed if ≥ PR achieved and no disease progression occurred within 60 days of last dose received
* Measurable disease
* Able to give voluntary written consent
* Eastern Cooperative Oncology Group performance status and/or other performance status 0, 1, or 2.
* Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3.
* Total bilirubin ≤ 1.5 × the upper limit of the normal range (ULN) (Total bilirubin ≥ 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.
* eGFR ≥ 20 mL/min/1.73 m2 (as calculated by Modified Diet in Renal Disease (MDRD) formula)

Exclusion Criteria:

* Non-AL amyloidosis
* Clinically overt myeloma
* Prior exposure to non-daratumumab anti-CD38 monoclonal antibodies.
* Clinically significant cardiac disease
* Severe obstructive airway disease
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Planned high-dose chemotherapy and autologous stem cell transplantation within 6, 28-day treatment cycles after starting on treatment.
* Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment.
* Infection requiring systemic intravenous antibiotic therapy or other serious infection within 14 days before study enrollment. Systemic treatment, within 14 days before the first dose, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, see Appendix 11.7), or use of Ginkgo biloba or St. John's wort.
* Positive for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Overall Complete Hematologic Response | Follow-up for up to 1 year
  Overall complete hematologic response rate will be defined as percentage of participants who achieve Complete Hematologic Response

SECONDARY OUTCOMES:
Duration of Very Good Partial Response (VGPR) or better hematologic response rates | Follow-up for up to 5 years
  Duration of hematologic VGPR or better response is defined as the time between the date of initial documentation of hematologic VGPR or better response to the date of first documented evidence of hematologic progressive disease.
Low-dFLC Partial Response Rate (applicable to low-dFLC pt group) | Follow-up for up to 1 year
  Percentage of participants who achieve a low-dFLC partial hematologic response rate and met criteria at screening for low-dFLC response assessment
Percentage of participants with an Organ Response | Follow-up for up to 3 years
  Organ response rate (OrRR) for kidney and cardiac is defined as the proportion of baseline organ involved participants who achieve organ response in each corresponding organ. Organ response defined for cardiac: N-terminal brain pronatriuretic peptide (NT-proBNP) response (> 30% and > 300 nanogram per liter [ng/L] decrease in participants with baseline NT-proBNP >= 650 ng/L) or New York Heart Association (NYHA) class response (>= 2 class decrease in participants with baseline NYHA class 3 or 4); for kidney: decrease in proteinuria by >=30% or below 0.5 grams /24 hours without renal progression.
Median estimate of months that participants have Progression Free Survival | Follow-up for up to 5 years
  Median estimate calculated using the Kaplan-Meier methodology
Median number of months of participant's Overall Survival | Follow-up for up to 5 years
  Overall survival (OS) is measured from the date of enrollment to the date of the participant's death
Time to Complete Hematologic Response | Follow-up for up to 1 year
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met the criteria for hematologic complete response.
Time to Hematologic Progression | Follow-up for up to 5 years
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met the criteria for hematologic progression
Time until Next Treatment Therapy | Follow-up for up to 5 years
  Measured in months from the date of enrollment to the start date of subsequent treatment for AL amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Cara Rosenbaum, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Boston University Medical Center, Boston, Massachusetts
  - Weill Cornell Medicine - Multiple Myeloma Center, New York, New York
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke M, Nieto M. AL Amyloidosis: Current Treatment and Outcomes. Adv Hematol. 2025 Mar 3;2025:7280805. doi: 10.1155/ah/7280805. eCollection 2025. PMID 40226119